CLINICAL TRIAL: NCT01826552
Title: Multicenter, Randomized, Open Label, Parallel Group Study to Evaluate the Safety and Efficacy of Orsiro Hybrid Drug Eluting Stent
Brief Title: Comparison of the Angiographic Result of the Orsiro Hybrid Stent With Resolute Integrity Stent
Acronym: ORIENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Jeju National University Hospital (Other); Chungbuk National University Hospital (Other); SMG-SNU Boramae Medical Center (Other); Korea University (Other); Inje University (Other); Kyung Hee University Hospital at Gangdong (Other); Inha University Hospital (Other)
Responsible Party: Principal Investigator, Tae-Jin Youn, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT01826552
Record Dates: First submitted 2013-03-03; First posted 2013-04-08 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Artery Disease; Coronary Heart Disease; Stable Angina; Unstable Angina; ST-segment Elevation Myocardial Infarction; Non-ST-segment Elevation Myocardial Infarction
Keywords: Orsiro hybrid stent; Drug-eluting stent; Zotarolimus-eluting stent; Coronary heart disease; Cobalt chromium
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Angina, Stable; Angina, Unstable; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orsiro (Experimental): The Patient group who are treated with Osiro Hybrid Drug-Eluting Stent (Biotronik AG, Bulach, Switzeland)
  Interventions: Device: Osiro Hybrid Drug-Eluting Stent
- Resolute Integrity (Active Comparator): The Patient group who are treated with ② Resolute Integrity zotarolimus-eluting stent (Medtronic Cardiovascular, CA, Minnesota, USA)
  Interventions: Device: Resolute Integrity

INTERVENTIONS:
Device: Osiro Hybrid Drug-Eluting Stent — Osiro Hybrid Drug-Eluting Stent (Biotronik AG, Bulach, Switzeland)
  Arms: Orsiro
Device: Resolute Integrity — Resolute Integrity zotarolimus-eluting stent (Medtronic Cardiovascular, CA, Minnesota, USA)
  Arms: Resolute Integrity

SUMMARY:
The purpose of this multicenter, randomized, open label, parallel arm study whether the newest 3rd generation stent - Orsiro hybrid sirolimus-eluting stent is noninferior to the newest 2nd generation stent - Resolute Integrity zotarolimus-eluting stent in terms of 9 months in-stent late lumen loss. 345 Korean patients with a wide variety of coronary heart disease will be enrolled to this "all-comers" trial to give definite answer to the above hypothesis that is urgently needed.

DETAILED DESCRIPTION:
The rate of restenosis after percutaneous coronary intervention (PCI) has dramatically decreased since the introduction of drug-eluting stents (DES). However, restenosis still remains a problem and some papers reported that the rate of restenosis can even go up to nearly 20% after the first-generation DES implantation, depending on the complexity of target lesion. Furthermore, there arises a concern about thrombogenic risk of these DES at the expense of reduced restenosis. Therefore, works aiming to reduce both restenosis and thrombosis are on-going, and there has been a rush of various second-generation DES with "biocompatible but non-absorbable polymer" and third-generation DES with "bioabsorbable polymer".

Recently, Orsiro hybrid sirolimus-eluting stent (Orsiro SES, Biotronik AG, Bulach, Switzeland) has been developed. It has a unique hybrid combination of polymers coated on thin cobalt-chromium struts (60um). The BIOlute® active component is a bioabsorbable polymer matrix combined with an anti-proliferative drug, sirolimus, and elutes the drug in a controlled manner after implantation, degrades over time and leaves only the PROBIO® coated stent behind in the long-term. The PROBIO® passive coating encapsulates the stent and protects interaction between the metal stent and the surrounding tissue. Although Orsiro SES showed excellent results in terms of late lumen loss at 9 months in first-in-man single arm trial (BIOFLOW-I trial), randomized controlled trials evaluating its efficacy and safety are limited to date.

The ORIENT Trial will evaluate the angiographic and clinical outcomes of the innovative third-generation DES, Orsiro SES, compared with the latest second-generation DES, Resolute Integrity zotarolimus-eluting stent (ZES-I, Medtronic Cardiovascular, Santa Rosa, California, USA), for treatment of patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the Orsiro Hybrid DES® or Endeavor Resolute Integrity® stent.
* He/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, acute myocardial infarction, recent infarction, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia) with a coronary artery or graft vessel lesion with >50% stenosis by visual estimation or >70% stenosis irrespective of the functional status.
* Target lesion(s) must be located in a coronary artery with estimated reference diameter of ≥ 2.5 mm and ≤ 5.0 mm.
* Target lesion(s) must be amenable for PCI.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Sirolimus, Zotarolimus, Cobalt chromium, Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.)
* Patients who cannot maintain aspirin, plavix from the study enrollment to study completion (during 1 year).
* Systemic (intravenous) Sirolimus or Zotarolimus use within 12 months.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or refuses blood transfusions.
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* Planned major non-cardiac surgery within the study period.
* Patients in cardiogenic shock
* Patients with symptomatic heart failure that preclude coronary angiography in supine position.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Late lumen loss (in-stent) | at 9 months
  Difference between the postprocedure and 9-month follow-up in-stent minimum lumen diameter. All QCA measurements of the target lesion will be obtained in the in-stent zone, and over entire segment including the stent and its 5 mm proximal and distal margins (in-segment zone).

SECONDARY OUTCOMES:
All-cause death | at 12 months
  All-cause mortality at 12 months follow-up
Cardiac death | at 12 months
  Cardiac death at 12 months follow-up. Any death due to proximate cardiac cause (eg, MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
Target lesion revascularization | at 12 months
  Any target lesion revascularization (TLR), defined as repeat revascularization within the stented segment including 5 mm proximal and distal border zones.
  TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLRs should be classified prospectively as clinically indicated* or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Target vessel revascularization | at 12 months
  Target vessel revascularization, defined as any revascularization of treated vessel.
  TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
Target-vessel related myocardial infarction | at 12 months
  Myocardial infarction (MI) was defined according to the ARC definitions and an extended historical protocol definition.
  Target vessel related MI is defined as MI, which developed in previously treated vessel.
Non-target vessel related myocardial infarction | at 12 months
  Myocardial infarction (MI) was defined according to the ARC definitions and an extended historical protocol definition.
  Non-target vessel related myocardial infarction is defined as MI, which developed in non-target vessel.
Clinical device success | Baseline
  Clinical Device Success is defined as an achievement of a final residual diameter stenosis of < 30% at the in-stent segment by online quantitative angiography or visual estimation, without device failure or malfunction. A device is considered to have failed if it did not meet the requirements of the definition for clinical device success.
Clinical lesion success | Baseline
  Clinical Lesion Success is defined as an achievement of a final in-stent segment diameter stenosis < 30% by online QCA or visual assessment over the entire stent length, with TIMI-3 flow and no more than an NHLBI type C dissection in the analysis segment
Clinical procedure success | Baseline
  Clinical Procedure Success is defined as an achievement of a final in-stent segment diameter stenosis < 30% by online QCA or visual assessment over the entire intervened vessel segment, with TIMI-3 flow and no more than an NHLBI type C dissection with or without any adjunctive devices, and without the occurrence of cardiac death, target vessel MI (Q-wave and non Q-wave MI), or repeat revascularization of the target lesion during the health care facility stay.
Stent thrombosis | at 12 months
  ARC definition of stent thrombosis is classified and defined as follows. Definite/Confirmed stent thrombosis refers angiographic or pathologic confirmation of partial or total thrombotic occlusion within the per-stent region with either i) acute ischemic symptoms, ii) ischemic EKG changes, iii) elevated cardiac biomarkers. Probable stent thrombosis is defined as any unexplained death within 30 days of stent implantation or any myocardial infarction, which is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause. Possible stent thrombosis is defined as any unexplained death beyond 30 days of stent implantation.
Target lesion failure | at 12 months
  Target lesion failure defined as a composite of cardiac death, myocardial infarction (not clearly attributed to a nontarget vessel), or clinically indicated target lesion revascularization by percutaneous or surgical methods at 1 years.
Patient-oriented composite outcome | at 12 months
  Patient-oriented composite outcome included all-cause mortality, any MI (including nontarget vessel territory), and any revascularization (including all target and nontarget vessels, regardless of percutaneous or surgical methods).
In-stent/in-segment % diameter stenosis | at 9 months
  Percent diameter stenosis in the in-stent and in-segment zone.
  All QCA measurements of the target lesion will be obtained in the in-stent zone, and over entire segment including the stent and its 5 mm proximal and distal margins (in-segment zone).
In-stent/in-segment binary restenosis | at 9 months
  Binary restenosis is defined as stenosis of 50% or more at follow-up angiography). All QCA measurements of the target lesion will be obtained in the in-stent zone, and over entire segment including the stent and its 5 mm proximal and distal margins (in-segment zone).
Clinically driven revascularization | at 12 months
  Clinically driven revascularization is considered clinically indicated if angiography at follow-up shows a percent diameter stenosis ≥ 50% (core laboratory quantitative coronary angiography assessment) and if one of the following occurs: (1) A positive history of recurrent angina pectoris, presumably related to the target vessel; (2) Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel; (3) Abnormal results of any invasive functional diagnostic test (eg, Doppler flow velocity reserve, fractional flow reserve); (4) A TLR or TVR with a diameter stenosis ≥ 70% even in the absence of the above-mentioned ischemic signs or symptoms.
Late lumen loss (in-segment) | at 9 months
  Difference between the postprocedure and 9-month follow-up in-segment minimum lumen diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Jin Youn, MD,PhD, Principal Investigator — Division of Cardiology, Department of Internal Medicine, College of Medicine, Seoul National University and Cardiovascular Center, Seoul National University Bundang Hospital; Dong-Ju Choi, MD,PhD, Study Chair — Division of Cardiology, Department of Internal Medicine and Cardiovascular Center, Seoul National University Bundang Hospital; In-Ho Chae, MD,PhD, Study Director — Division of Cardiology, Department of Internal Medicine and Cardiovascular Center, Seoul National University Bundang Hospital
Locations (8):
- South Korea (8):
  - Korea University Ansan Hospital, Ansan
  - Chungbuk University Hospital, Cheongju-si
  - Inje University Ilsan Paik Hospital, Ilsan
  - Inha University Hospital, Incheon
  - Jeju University Hospital, Jeju City
  - Seoul National University Bundang Hospital, Seongnam
  - Boramae Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong Hospital, Seoul

REFERENCES:
- [Derived] Lee JM, Park SD, Lim SY, Doh JH, Cho JM, Kim KS, Bae JW, Chung WY, Youn TJ. Angiographic and clinical comparison of novel Orsiro Hybrid sirolimus-eluting stents and Resolute Integrity zotarolimus-eluting stents in all-comers with coronary artery disease (ORIENT trial): study protocol for a randomized controlled trial. Trials. 2013 Nov 20;14:398. doi: 10.1186/1745-6215-14-398. PMID 24257456